CLINICAL TRIAL: NCT00667927
Title: Autologous Bone Marrow Transplant for Children With AML in First Complete Remission: Use of Marker Genes to Investigate the Biology of Marrow Reconstitution and the Mechanism of Relapse
Brief Title: Autologous Bone Marrow Transplant for Children With Acute Myelogenous Leukemia (AML) in First Complete Remission
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Hale, Gregory A, St. Jude Children's Research Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMLREM
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Last update posted 2008-04-28 (Estimated); Status verified 2008-04

CONDITIONS: Acute Myeloid Leukemia
Keywords: Autologous bone marrow transplant; gene marking
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Busulfan; Cyclophosphamide; Mesna

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Drug: Busulfan; Drug: Cyclophosphamide; Drug: Mesna

INTERVENTIONS:
Drug: Busulfan — See Detailed Description section for description of treatment plan.
  Other Names: Myleran
Drug: Cyclophosphamide — See Detailed Description section for description of treatment plan.
  Other Names: Cytoxan, CTX
Drug: Mesna — See Detailed Description section for description of treatment plan.
  Other Names: MESNCX

SUMMARY:
This study proposes to transfer marker genes (detectable genetic traits or segments of DNA that can be identified and tracked) into aliquots of marrow obtained for Bone Marrow Transplant (BTM) in patients in remission of Acute Myelogenous Leukemia (AML).

DETAILED DESCRIPTION:
The primary objective of this study was to estimate the continuous complete remission rate at 2 years post transplant for children with AML in first complete remission treated with autologous BMT.

Secondary objectives used transduction of marker genes into autologous marrow to determine the following:

1. whether the source of relapse after BMT for AML is residual malignant cells in the harvested marrow or in the patient, and whether marrow purging is therefore rational.
2. whether the majority of AML, which lack genetic markers, represent abnormalities in a multi-lineage progenitor cell, and whether therefore, auto grafting/intensified chemotherapy is ever likely to augment the cure rate.
3. the mechanisms of autologous reconstitution, and the effects of stimuli which modify the process.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 1 and 18 years at diagnosis with acute nonlymphocytic leukemia in first remission are eligible for this protocol.
* Patients enrolled on the AML-87 study in second or subsequent remission are eligible for this protocol.

Exclusion Criteria:

* Has an HLA-matched, MLC-compatible donor(unless parents and/or patient refuses transplant.
* Diagnosis of FAB M3 or FAB M3v (acute progranulocytic leukemia)
* Life expectancy limited by disease other than leukemia
* Significant cardiac disease (echo shortening fraction <25% or MUGA scan <50%)
* Severe renal dysfunction, i.e., creatinine clearance less than 60cc/1.73 m2/min
* Severe restrictive pulmonary disease (FCV less than 40% of predicted)
* Severe hepatic disease (bilirubin greater than 3 mg/dl or SGPT greater than 500IU)
* Severe personality disorder or mental illness
* Previous severe cystitis from cyclophosphamide
* Previous total dose of anthracyclines of >450 mg/m2
* Sever infection that on evaluation by the PI precludes ablative chemotherapy or successful transplantation
* Previous autologous transplant
* HIV reactivity
* Karnofsky score <70%

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 1991-03; Primary Completion 1995-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
To estimate the continuous complete remission rate at 2 years for children with AML in first complete remission treated with Autologous Bone Marrow Transplant (ABMT). | 2 years post transplant

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A Hale, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: Related Info — http://www.stjude.org